CLINICAL TRIAL: NCT01559844
Title: An Open-Label Study to Explore the Clinical Efficacy of GS-7977 With Ribavirin Administered Pre-Transplant in Preventing Hepatitis C Virus (HCV) Recurrence Post-Transplant
Brief Title: Efficacy of Sofosbuvir With Ribavirin Administered Pre-Transplant in Preventing Hepatitis C Virus (HCV) Recurrence Post-Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P7977-2025
Record Dates: First submitted 2012-03-05; First posted 2012-03-21 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-06

CONDITIONS: Hepatitis C; Hepatocellular Carcinoma
Keywords: Hepatitis; Chronic; hepatocellular carcinoma; HCC; transplant
MeSH Terms: conditions — Hepatitis C; Carcinoma, Hepatocellular; Hepatitis; Bronchiolitis Obliterans Syndrome | interventions — Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SOF+RBV (Experimental): Sofosbuvir plus ribavirin for up to 48 weeks or until time of transplant, whichever occurs first.
  Interventions: Drug: Sofosbuvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir 400 mg (2 x 200 mg tablets) administered orally once daily
  Other Names: GS-7977; PSI-7977; Sovaldi®
Drug: Ribavirin — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg)

SUMMARY:
The primary objective is to determine if the administration of a combination of sofosbuvir (SOF; GS-7977; PSI-7977) and ribavirin (RBV) to HCV-infected adults with hepatocellular carcinoma (HCC) meeting the MILAN criteria prior to undergoing liver transplantation could prevent post-transplant re-infection as determined by a sustained post-transplant virological response (HCV RNA < LLoQ) at 12 weeks post-transplant.

Participants will enroll in the pretransplant treatment phase (24 or 48 weeks). Participants enrolling for 24 weeks in the pretransplant treatment phase may receive treatment for up to an additional 24 weeks in the pretransplant retreatment phase. Participants enrolling for 48 weeks in the pretransplant treatment will have a second baseline at Week 24 for combined analysis in the pretransplant retreatment phase.

Participants who undergo liver transplant will stop all study drug 24 hours prior to transplant, and enter a 48-week follow-up phase to monitor for recurrent HCV infection.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Males or females, age > 18 years old
3. Males must agree to consistently and correctly use a condom while their female partner agrees to use an approved form of birth control from the date of screening until 7 months after their last dose of ribavirin.
4. Confirmation of chronic HCV infection documented by at least one measurement of serum HCV RNA above the LLOQ measured at screening, and at least one of the following:

   * Positive anti-HCV antibody test, HCV RNA or HCV genotyping test at least 6 months prior to the baseline/Day 1 visit together with positive HCV RNA test and anti-HCV antibody at the time of screening, or
   * Positive HCV RNA test and anti-HCV antibody test at the time of screening together with either a liver biopsy consistent with chronic HCV infection (or a liver biopsy performed before enrollment with evidence of chronic HCV infection, such as the presence of fibrosis)
5. HCV RNA > 10^4 IU/mL at screening
6. Patients meeting the MILAN criteria undergoing liver transplant for HCC secondary to HCV with a MELD of < 22 and a HCC weighted MELD of ≥ 22.
7. Child-Pugh Score (CPT) ≤ 7
8. Planned management of the subject to meet United Network for Organ Sharing (UNOS) criteria, with imaging studies made available for review if required.
9. Has not been treated with any investigational drug or device within 30 days of the screening visit.

Exclusion Criteria:

1. Females of child-bearing potential who is pregnant or nursing
2. Prior exposure to a direct-acting antiviral targeting the HCV nonstructural (NS)5B polymerase
3. Any transplant patient who has agreed to a liver transplant from a live donor.
4. Participants requiring planned induction therapy with biologics posttransplantation or with a posttransplantation immunosuppressive regimen not consistent with the following within the first 12 weeks posttransplant:

   * Solumedrol/Prednisone (tapering over approximately 7 days)
   * Tacrolimus (maintaining a serum level of 5 12 ng/mL)
   * Mycophenolate mofetil (up to 2 g/day)
   * Introduction of new maintenance immunosuppressants different from the above list is disallowed except in consultation during the first 12 weeks posttransplant
5. Current, uncontrolled ascites, variceal hemorrhage, hepatic encephalopathy, hepatorenal syndrome and hepatopulmonary syndrome, among other signs of decompensated cirrhosis.
6. Chronic liver disease of a non-HCV etiology (eg, hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, cholangitis)
7. Infection with hepatitis B virus (HBV) or HIV
8. Contraindications to RBV therapy
9. Chronic use of systemically administered immunosuppressive agents (eg, prednisone equivalent > 10 mg/day) in the pretransplant treatment period.
10. History of previous solid organ transplantation
11. Evidence of renal impairment (CLcr < 60 mL/min) calculated by the Cockcroft-Gault equation.
12. History or current evidence of psychiatric illness, immunologic disorder, hemoglobinopathy, pulmonary or cardiac disease, porphyria, or poorly controlled diabetes, cancer other than HCC, or a history of malignancy that in the opinion of the investigator makes the patient unsuitable for the study. Patients with clinical signs or symptoms of acute pancreatitis with elevated lipase (at Screening or during the screening period)
13. Known hypersensitivity to RBV, the study investigational medicinal product, the metabolites, or formulation excipients
14. History of having received any systemic antineoplastic (including sorafenib) or immunomodulatory treatment (including radiation) within 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study (excluding a local regional therapy such as TACE).
15. Treatment with Transcatheter arterial chemoembolization (TACE) or radio frequency ablation (RFA) within 30 days prior to the first dose.
16. Participation in a clinical study with an investigational drug, biologic, or device within 3 months prior to first dose administration at the baseline/Day 1 Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Denning, MA, Study Director — Gilead Sciences
Locations (15):
- United States (13):
  - UCLA Medical Center-The Pfleger Liver Institute, Los Angeles, California
  - UC San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - St. Louis University Hospital, St Louis, Missouri
  - Columbia University, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Baylor Health Care System, Dallas, Texas
- Auckland Clinical Studies, Auckland, New Zealand
- Liver Unit Clinica University de Navara, Pamplona, Spain

REFERENCES:
- [Derived] Babusis D, Curry MP, Kirby B, Park Y, Murakami E, Wang T, Mathias A, Afdhal N, McHutchison JG, Ray AS. Sofosbuvir and Ribavirin Liver Pharmacokinetics in Patients Infected with Hepatitis C Virus. Antimicrob Agents Chemother. 2018 Apr 26;62(5):e02587-17. doi: 10.1128/AAC.02587-17. Print 2018 May. PMID 29439971
- [Derived] Curry MP, Forns X, Chung RT, Terrault NA, Brown R Jr, Fenkel JM, Gordon F, O'Leary J, Kuo A, Schiano T, Everson G, Schiff E, Befeler A, Gane E, Saab S, McHutchison JG, Subramanian GM, Symonds WT, Denning J, McNair L, Arterburn S, Svarovskaia E, Moonka D, Afdhal N. Sofosbuvir and ribavirin prevent recurrence of HCV infection after liver transplantation: an open-label study. Gastroenterology. 2015 Jan;148(1):100-107.e1. doi: 10.1053/j.gastro.2014.09.023. Epub 2014 Sep 28. PMID 25261839

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Spain, and New Zealand. The first participant was screened on 27 March 2012. The last study visit occurred on 20 October 2014.
Pre-assignment Details: 92 participants were screened.
Groups:
- SOF+RBV: Sofosbuvir (SOF) 400 mg tablet once daily + ribavirin (RBV) tablets (1000-1200 mg daily based on weight) for up to 48 weeks or until time of transplant, whichever occured first.
Period: Overall Study
Arm/Group | SOF+RBV
Started | 61
Completed | 36
Not Completed | 25
Not completed — Consent Withdrawn | 7
Not completed — Death | 5
Not completed — Efficacy Failure | 10
Not completed — No Longer A Transplant Candidate | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were enrolled and received at least 1 dose of study drug
Groups:
- SOF+RBV: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for up to 48 weeks or until time of transplant, whichever occured first.
Arm/Group | SOF+RBV
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 55
  Black or African American | 6
Region of Enrollment [Number; unit: participants]
  United States | 55
  Spain | 5
  New Zealand | 1
Prior Hepatitis C Virus (HCV) Treatment [Number; unit: participants]
  Yes | 46
  No | 15
Response to Last Prior HCV Treatment Regimen [Number; unit: participants]
  Non-Responder: Null | 11
  Non-Responder: Partial | 11
  Responder: Breakthrough | 3
  Responder: Relapser | 9
  Unknown | 12
  Had Not Received Prior Treatment | 15
Days on Transplant Waitlist [Mean (Standard Deviation); unit: days] | 266 (488.8)
Baseline HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.14 (0.633)
Baseline HCV RNA Category [Number; unit: participants]
  < 6 log10 IU/mL | 20
  ≥ 6 and < 7 log10 IU/mL | 38
  ≥ 7 log10 IU/mL | 3
HCV Genotype [Number; unit: participants] — There are variations of HCV which are all similar enough to be called HCV, but are distinct enough to be referred to as HCV genotypes.
  participants
    Genotype 1a | 24
    Genotype 1b | 21
    Genotype 2a | 1
    Genotype 2b | 7
    Genotype 3a | 7
    Genotype 4a | 1
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 13
    CT | 39
    TT | 8
    Missing | 1
Baseline Child-Pugh Turcotte (CPT) Score [Number; unit: participants] — CPT scores, widely used to grade the severity of cirrhosis and to determine the need for liver transplantation, are calculated based on a combination of laboratory values and clinical features. CPT scores can range from 5 to 15, with higher scores indicating a greater severity of disease.
  participants
    5 | 26
    6 | 18
    7 | 14
    8 | 3
Baseline Model For End-Stage Liver Disease (MELD) Score [Number; unit: participants] — MELD scores, used to assess prognosis and suitability for transplant, are calculated based on laboratory values only and can range from 6 to 40, with higher scores indicating greater disease severity.
  participants
    6 | 5
    7 | 18
    8 | 12
    9 | 9
    10 | 6
    11 | 8
    13 | 2
    14 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Posttransplant Virologic Response (pTVR) at Posttransplant Week 12
Description: pTVR was defined as HCV RNA < the lower limit of quantification (LLOQ, ie, 25 mL/IU) at Week 12 after transplant.
Time Frame: Posttransplant Week 12
Population: Participants in the Full Analysis Set (enrolled and received at least 1 dose of study drug) who underwent liver transplantation, and who had HCV RNA < LLOQ at last measurement prior to transplant were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV
Number analyzed (Participants) | 43
percentage of participants
  Transplant after ≥ 12 weeks of treatment (N=32) | 75.0
  Transplant after any duration of treatment (N=43) | 69.8

2. Primary Outcome: Percentage of Participants Experiencing Any Adverse Event Leading to Permanent Discontinuation of Sofosbuvir Prior to Receiving Transplant
Time Frame: Up to 48 weeks prior to transplant
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV
Number analyzed (Participants) | 61
percentage of participants | 3.3

3. Primary Outcome: Percentage of Participants With Graft Loss Following Transplant
Time Frame: Up to 48 weeks following transplant
Population: Participants in the Safety Analysis Set who underwent liver transplantation were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV
Number analyzed (Participants) | 46
percentage of participants | 6.5

4. Secondary Outcome: Percentage of Participants With Posttransplant Virologic Response (pTVR) Through Posttransplant Week 48
Description: pTVR was defined as HCV RNA < the lower limit of quantification (LLOQ, ie, 25 mL/IU) at the relevant time point after transplant.
Time Frame: Up to 48 weeks following transplant
Population: Participants in the Full Analysis Set who underwent liver transplantation and who had ≥ 12 weeks treatment and HCV RNA < LLOQ at last measurement prior to transplant were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV
Number analyzed (Participants) | 32
percentage of participants
  Posttransplant Week 1 (N = 32) | 87.5
  Posttransplant Week 2 (N = 32) | 81.3
  Posttransplant Week 4 (N = 32) | 75.0
  Posttransplant Week 8 (N = 32) | 75.0
  Posttransplant Week 24 (N = 32) | 75.0
  Posttransplant Week 48 (N = 30) | 66.7

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ (ie, 25 mL/IU) During Treatment Through Week 48
Time Frame: Up to 48 weeks prior to transplant
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV
Number analyzed (Participants) | 61
percentage of participants
  Week 1 (N = 61) | 13.1
  Week 2 (N = 61) | 57.4
  Week 3 (N = 60) | 81.7
  Week 4 (N = 58) | 93.1
  Week 8 (N = 54) | 90.7
  Week 12 (N = 48) | 93.8
  Week 24 (N = 30) | 100.0
  Week 36 (N = 9) | 100.0
  Week 48 (N = 8) | 100.0

6. Secondary Outcome: HCV RNA and Change From Baseline in HCV RNA Through Week 8
Time Frame: Up to 8 weeks prior to transplant
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF+RBV
Number analyzed (Participants) | 61
log10 IU/mL
  Week 1 (N = 59) | -3.87 (0.700)
  Week 2 (N = 61) | -4.43 (0.771)
  Week 3 (N = 60) | -4.64 (0.670)
  Week 4 (N = 58) | -4.69 (0.686)
  Week 8 (N = 53) | -4.66 (0.708)

7. Secondary Outcome: Proportion of Participants With Virologic Failure Prior to Transplant
Description: Virologic failure (VF) in the pretransplant phase was defined by:
  * Breakthrough (HCV RNA ≥ 25 IU/ml after having previously had HCV RNA < 25 IU/ml, while on treatment)
  * Rebound (breakthrough or > 1 log10 IU/ml increase in HCV RNA from nadir while on treatment)
  * Non-response (HCV RNA ≥ 25 IU/ml through 8 weeks of treatment)
  * Pre-transplant relapse (HCV RNA ≥ 25 IU/ml during the Pre-Transplant off-treatment follow-up period after having achieved HCV RNA < 25 IU/ml at last observed HCV RNA on treatment)
Time Frame: Up to 48 weeks prior to transplant
Population: On-treatment VF: Full Analysis Set. Posttreatment/Pretransplant VF - 24 Weeks or 48 Weeks: Participants who completed 24 or 48 weeks of treatment and had an observed or imputed Week 4 posttreatment follow-up HCV RNA value relapsed during posttreatment follow-up were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV
Number analyzed (Participants) | 61
percentage of participants
  On-treatment VF (N = 61) | 8.2
  Posttreatment/Pretransplant VF - 24 Weeks (N = 15) | 73.3
  Posttreatment/Pretransplant VF - 48 Weeks (N = 8) | 37.5

8. Primary Outcome: Number of Participants Who Died
Description: * Treatment-emergent deaths were those that occurred while taking study drug or to the minimum of 1) date of transplantation, 2) retreatment 1st dose date, or 3) last dose date + 30 days.
  * Only those participants who underwent liver transplantation were analyzed for death post-transplantation.
Time Frame: Up to 48 weeks following transplant
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | SOF+RBV
Number analyzed (Participants) | 61
participants
  All Deaths | 5
  Treatment-Emergent Death (N = 61) | 1
  Death Following Transplant (N = 46) | 3
  Death Not Meeting Either Criteria (N = 61) | 1

ADVERSE EVENTS:
Time Frame: Up to 48 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF+RBV
Serious Adverse Events (participants affected / at risk) | 11/61
Other Adverse Events (participants affected / at risk) | 49/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV (N=61)
Atrial fibrillation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 1
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Cellulitis (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Peritonitis bacterial (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV (N=61)
Anaemia (Blood and lymphatic system disorders) | 13
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 10
Fatigue (General disorders) | 23
Oedema peripheral (General disorders) | 4
Urinary tract infection (Infections and infestations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 4
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 14
Insomnia (Psychiatric disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years